CLINICAL TRIAL: NCT00616200
Title: The Effect of a Very Low Carbohydrate Diet on Symptoms of Irritable Bowel Syndrome: A Prospective Pilot Study
Brief Title: Effects of a Very Low Carbohydrate Diet on Symptoms of Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-2899; GCRC 2392
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2011-10

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome
Keywords: D-IBS (diarrhea predominant irritable bowel syndrome)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Other: Very low carbohydrate diet

INTERVENTIONS:
Other: Very low carbohydrate diet — 4 weeks on strictly controlled low carbohydrate diet

SUMMARY:
The purposes of this study are to prospectively determine the effect of a very low carbohydrate diet on quality of life and gastrointestinal symptoms in patients with diarrhea-predominant irritable bowel syndrome (IBS-D); and to determine possible physiological correlates of symptom improvement, as related to post-prandial 5-hydroxytryptamine (5-HT) release, weight loss and fiber content.

DETAILED DESCRIPTION:
Approximately 10-15% of individuals in the United States have symptoms consistent with irritable bowel syndrome (IBS) which is a costly disorder and negatively impacts patient quality of life. The pathogenesis of this heterogeneous disorder is still not well understood. Patients frequently identify worsening of symptoms after meals and often cite particular foods as triggers of their IBS symptoms. Unfortunately, there is insufficient randomized clinical trial data to allow for specific dietary recommendations. Previous research has suggested a role for carbohydrate ingestion in IBS. There is also evidence for the role of the post-prandial release of 5-hydroxytryptamine (5-HT) and its turnover (as represented by the ratio of its metabolite, 5-hydroxyindoleacetic acid (5-HIAA), to 5-HT in response to a carbohydrate-rich meal, especially in those with IBS-D. As the prevalence of overweight (body mass index [BMI] > 25 kg/m2) and obesity (BMI > 30 kg/m2) has risen in recent years, very low carbohydrate diets have become popular for those attempting to lose weight. Patients with IBS, especially IBS-D, anecdotally report improvement in their gastrointestinal symptoms after initiating a very low carbohydrate diet. However, no study has investigated the effect of a very low carbohydrate diet on symptoms and quality of life in patients with IBS-D.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, male or female
2. Meet Rome II Criteria for IBS-D
3. Body mass index > 25 kg/m^2
4. Desire to use a very low carbohydrate diet for weight loss
5. Score of > 36 on the FBDSI
6. Ability to understand consent form
7. In stable health by screening history, physical examination performed by a study physician, laboratory tests (normal blood counts, kidney function tests, liver tests, TSH).

Exclusion Criteria:

1. Age < 18 years or age > 70 years
2. History of inflammatory bowel disease
3. History of any gastrointestinal surgery that preceded the onset of IBS symptoms
4. Pregnancy or breastfeeding
5. FBDSI symptom score of ≤ 36
6. Inability to understand consent form
7. Diabetes requiring medications (must be controlled with diet and exercise alone).
8. Chronic narcotic use for any reason
9. Use of serotonin-selective reuptake inhibitors unless patient has been on a stable dose for at least 4 weeks.
10. Use of any over-the-counter or prescription weight loss medications.
11. Any chronic or unstable diseases (e.g., kidney disease, heart disease, or cancer) that may put the subject at increased risk from the intervention
12. Any of the following baseline abnormalities of laboratory tests or physical exam findings:

    1. Serum creatinine > 1.5 mg/dL in men, > 1.3 mg/dL in women.
    2. Liver disease (AST or ALT > 2 times the upper limit of normal or total bilirubin > 1.6mg/dL).
    3. Blood pressure > 160/100 mm Hg.
    4. Fasting triglycerides > 600 mg/dL.
    5. Fasting serum low-density lipoprotein (LDL) cholesterol > 190 mg/dL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Drossman, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Center for Functional GI & Motility Disorders, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Austin GL, Dalton CB, Hu Y, Morris CB, Hankins J, Weinland SR, Westman EC, Yancy WS Jr, Drossman DA. A very low-carbohydrate diet improves symptoms and quality of life in diarrhea-predominant irritable bowel syndrome. Clin Gastroenterol Hepatol. 2009 Jun;7(6):706-708.e1. doi: 10.1016/j.cgh.2009.02.023. Epub 2009 Mar 10. PMID 19281859

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients responded to advertising in local media for participation in a research study looking at IBS-D. Patients presented to the General Clinical Research Center at the University of North Carolina. Each of the six weekly study visits and one baseline visit was conducted at the UNC GCRC.
Groups:
- Standard Diet Then Very Low Carbohydrate Diet: Two weeks of a carbohydrate rich diet was followed by four weeks of A Very Low Carbohydrate Diet. VLCD = <20g/day of carbohydrates
Period: Two Week Standard Diet
Arm/Group | Standard Diet Then Very Low Carbohydrate Diet
Started | 17
Completed | 16
Not Completed | 1
Period: Four Week Very Low Carbohydrate Diet
Arm/Group | Standard Diet Then Very Low Carbohydrate Diet
Started | 16
Completed | 13
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Four Week Very Low Carbohydrate Diet: A Very Low Carbohydrate Diet was administered for four weeks. VLCD = <20g/day of carbohydrates
Arm/Group | Four Week Very Low Carbohydrate Diet
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 2
Region of Enrollment [Number; unit: participants]
  North America | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting "Adequate Relief" From IBS Symptoms for the Previous Week. Adequate Relief Was a "True/False" Item.
Description: Adequate relief was measured as the primary endpoint via a single item Adequate Relief Question asking "Over the past week have you had adequate relief of your symptom experience". Higher scores represent greater levels of adequate relief over the week prior to the assessment. Participants completed this 1-item questionnaire at the end of each of weeks of the study, assessing whether they had adequate relief of their IBS symptoms for the week.
  A responder was defined as reporting adequate relief in at least 2 of the 4 weeks on the VLCD.
Time Frame: At the end of each of 6 study weeks
Measure: Number; unit: Participants
Arm/Group | Four Week Very Low Carbohydrate Diet
Number analyzed (Participants) | 17
Participants | 13

2. Secondary Outcome: Impact of Very Low Carbohydrate Diet on Stool Frequency
Description: Stool Frequency was measured as number of stools per day
Time Frame: 6 Weeks
Population: Analysis was per protocol analysis
Measure: Mean (Standard Deviation); unit: Stools Per day
Arm/Group | Four Week Very Low Carbohydrate Diet
Number analyzed (Participants) | 17
Stools Per day | 2.6 (.8)

3. Secondary Outcome: Sickness Impact Profile
Description: Units of measurement on the Sickness Impact Profile were ordinal rated scored. Information on scoring use and interpretation of the Sickness Impact Profile, readers are encouraged to read Bergner et. al. 1981 - Bergner, M., Bobbit, R.A., Carter, W.B. et all (1981) the Sickness Impact Profile: Development and final revision of a health status measure. Medical Care, 19:787-805 The SIP measures sickness-related dysfunction based on behavior in order to provide a measure of health status that will aid in assessing the outcome of health care services.
Time Frame: At the end of four week VLCD
Population: The scoring range is from no impairment with a score of 0, to significant impairment, with 5. Changes in score of 3.5 are considered clinically significant.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Four Week Very Low Carbohydrate Diet
Number analyzed (Participants) | 17
Scores on a scale | 2.3 (3.6)
Statistical Analysis 1: Comparison: Four Week Very Low Carbohydrate Diet; Sickness Impact Profile scores improved; Test type: Superiority or Other; p = .001, ANOVA

ADVERSE EVENTS:
Arm/Group | Four Week Very Low Carbohydrate Diet
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
Low N, lack of standard control group and specific overweight/obese female predominant population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes